CLINICAL TRIAL: NCT01212497
Title: Virtual Coach for Mindfulness Meditation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychometrix Associates (Industry)
Responsible Party: Dr. Eva Hudlicka, Psychometrix Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2010-09-30 (Estimated); Status verified 2010-09

CONDITIONS: Mindfulness Training
Keywords: mindfulness; meditation; training; coaching; virtual coach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness meditation coaching (Experimental): Assess effectiveness of using a virtual computer coach to train mindfulness meditation
  Interventions: Behavioral: Mindfulness meditation coaching

INTERVENTIONS:
Behavioral: Mindfulness meditation coaching — Participants interact with virtual coach to obtain instruction in mindfulness meditation and coaching support.

SUMMARY:
Evaluate the effectiveness of using a virtual computer coach to provide mindfulness meditation training, and the coaching support required to initiate a regular practice.

ELIGIBILITY:
Inclusion Criteria:

* over 18, no previous mindfulness experience, computer literacy

Exclusion Criteria:

* substance abuse, anxiety/depression, psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Frequency of meditating | 7 weeks (weekly)
  Measure the number of times participants meditated per week, throughout the 7 week period of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Hudlicka, Ph.D., Principal Investigator — Psychometrix Associates
Locations (1):
- Psychometrix Associates, Blacksburg, Virginia, United States